CLINICAL TRIAL: NCT03208764
Title: A Prospective, Open Labeled, Multi-Center, Evaluation of the Efficacy Safety and Tolerability of Nitric Oxide Given Intermittently Via Inhalation to Subjects With NTM (Specifically MABSC)
Brief Title: Inhaled Nitric Oxide for Patients With MABSC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beyond Air Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIT_ CP_ CFNTM_01
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2017-07

CONDITIONS: Mycobacterium Abscessus Infection
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nitric Oxide treatment (Experimental)
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Subjects will be treated with 91 thirty minute sessions of 160 ppm Nitric Oxide with at least 3 hours between each session.

SUMMARY:
A Prospective, Open labeled, multi-Center, Evaluation of the Efficacy Safety and Tolerability of Nitric Oxide Given Intermittently via Inhalation to Subjects with NTM (specifically MABSC)

Nitric Oxide (NO) has been shown to play a critical role in various biological functions. In the airways, NO is considered to play a key role in the innate immune system in which the first-line of host defense against microbes is built.

In vitro studies suggested that NO, in part per million (ppm) concentrations, possesses anti-microbial activity against a wide variety of phyla including fungi, and antibiotic-resistance bacteria.

In this study the investigators wish to evaluate the efficacy, safety and tolerability of 160 ppm Nitric Oxide intermittently delivered via inhalation to subjects infected with Non-tuberculosis mycobacteria (NTM), specifically with MABSC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (Male or female) between 6 to 65 years old
2. Diagnosis of pulmonary non-tuberculosis mycobacterial lung disease in accordance with the 2007 ATS/IDSA criteria with evidence of nodular bronchiectasis and/or cavitary disease by chest computed tomography (CT) and by culture.
3. History of at least 6 months chronic infection with Mycobacterium abscessus.
4. Mycobacterium abscessus positive sputum sample at screening or prior to screening.
5. Receiving ATS/IDSA guidelines-based treatment regimen defined as: adherent to a multi-drug regimen for at least 6 months prior to screening with persistently positive mycobacterial abscessus cultures.
6. FEV1 ≥ 30% at screening as well as baseline.
7. Ability to produce sputum or be willing to undergo an induction of sputum for clinical evaluation.
8. Life expectancy ≥1 year
9. Ability to perform 6MWT, but not to exceed a distance of 700 meters during screening.
10. Ability to understand and comply with study requirements.
11. Approved and signed informed consent by subject and/or by parent/legal guardian (depending on subject's age).

Exclusion Criteria:

1. Breastfeeding or pregnancy as evidenced by a positive pregnancy test.
2. Subjects diagnosed with methemoglobinemia, immunodeficiency, heart disease, pulmonary hypertension and/or high blood pressure.
3. Use of an investigational drug during the last 30 days prior enrollment and/or the subject is expected to participate in a new study within five months from enrollment to this study.
4. History of frequent epistaxis (>1 episode/month).
5. Significant hemoptysis during the last 30 days prior to enrolment (>30 Ml of blood in a 24-hour period).
6. Methemoglobin level >2% at screening.
7. Patients on inconsistant dosage of systemic steroids (any formulation) 30 days prior to enrolment.
8. History of illicit drug or medication abuse within 1 year of screening.
9. History of lung transplantation.
10. History of daily, continuous oxygen supplementation.
11. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data.
12. Pulmonary tuberculosis requiring treatment or treated within 2 years prior to screening.
13. Any change in chronic NTM multi-drug regimen within 28 days prior to study day 1.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Safety measured by NO-related Serious Adverse Events | 21 days

SECONDARY OUTCOMES:
Six minute walk test | 21 days
Mycobacterium Abscesuss load in sputum | 81 days
NO-related AE's such as elevation of methemoglobin and elevation of NO2 during treatment | 21 days
Type and frequency of occurrence of NO-related Adverse Events (AE's) and Serious AE's (SAE's) | 51 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel